CLINICAL TRIAL: NCT00226265
Title: The Short Form-36: Pre-vs. Post-Surgical Administration in Cardiac Surgery Patients
Brief Title: The Short Form-36: Pre- Versus Post-Surgical Administration in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary E. Charlson, MD, Principal Investigator, Weill Medical College of Cornell University
Other Study IDs: 1203-069
Record Dates: First submitted 2005-09-14; First posted 2005-09-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Bypass Grafting; Heart Diseases; Heart Valve Diseases
Keywords: Cardiac surgery patients; Quality of Life; Recall bias; Aortic valve replacement; Mitral valve replacement; Tricuspid valve replacement; Coronary artery bypass graft surgery
MeSH Terms: conditions — Heart Diseases; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether the SF-36 can be administered reliably to cardiac surgery patients (two to three days) post-surgery, with the patient answering the questions of this survey from a pre-surgical perspective.

DETAILED DESCRIPTION:
The purpose of this study, is to determine whether the SF-36 can be administered reliably to cardiac surgery patients (two to three days) post-surgery, with the patient answering the questions of this survey from a pre-surgical perspective.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery patients who are between the ages of 18 and 100
* Are English speaking
* Able to give consent
* Undergoing cardiac surgery including (but not limited to):

  * Aortic valve replacement (AVR)
  * Mitral valve replacement (MVR)
  * Tricuspid valve replacement (TVR)
  * Coronary artery bypass graft (CABG).

Exclusion Criteria:

* Non-cardiac surgery patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac Surgery Patients at New York Presbyterian Hospital-Weill Cornell Medical College
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 1999-01 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The New York Presbyterian Hospital-Weill Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No Plan to Share IPD